CLINICAL TRIAL: NCT00757341
Title: An Open-Label, Single-Dose Study of the Mass Balance and Metabolic Disposition of Orally Administered [14C]-Labeled Bosutinib in Healthy Male Subjects
Brief Title: Study Evaluating The Mass Balance And Metabolic Disposition Of SKI-606
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-1112-US
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SKI-606 (Experimental)
  Interventions: Drug: SKI-606

INTERVENTIONS:
Drug: SKI-606

SUMMARY:
This study will assess the mass balance, metabolic disposition, and identification of metabolites following single oral administration of [14C]-SKI-606 in healthy male subjects.

ELIGIBILITY:
Healthy men, aged 18 to 50 years.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mass Balance and Metabolic Disposition | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tacoma, Washington, United States